CLINICAL TRIAL: NCT01131039
Title: A Phase II Trial of Gemcitabine Plus Bevacizumab in Patients With Platinum-Resistant Ovarian, Primary Peritoneal or Fallopian Tube Cancer
Brief Title: Safety and Efficacy Study of Gemcitabine Plus Bevacizumab in Patients With Platinum-Resistant Ovarian, Primary Peritoneal or Fallopian Tube Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left Emory
Sponsor: Emory University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00023366; AVF4314S (Other: Other)
Record Dates: First submitted 2010-05-21; First posted 2010-05-26 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Fallopian Tube Neoplasms; Ovarian Cancer; Primary Peritoneal
Keywords: Ovarian Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Gemcitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single (Experimental)
  Interventions: Drug: Gemcitabine/Bevacizumab

INTERVENTIONS:
Drug: Gemcitabine/Bevacizumab — Gemcitabine: IV, days 1,8, and every 21 days
  Bevacizumab: IV, day 1 and every 21 days until disease progression
  Other Names: Gemcitabine; Gemzar®; Bevacizumab; Avastin

SUMMARY:
The purpose of the study is to determine whether the administration of bevacizumab and gemcitabine given by IV infusion can prolong survival, delay tumor growth, and/or shrink tumors in patients with ovarian cancer, primary peritoneal, or fallopian tube cancer.

ELIGIBILITY:
Inclusion Criteria:

Patients must have platinum-resistant ovarian, primary peritoneal or fallopian tube cancer.

Patients will be included in the study based on the following criteria:

1. Signed informed consent
2. Age ≥ 19 yrs
3. Advanced, histologically documented ovarian, primary peritoneal, or fallopian tube cancer
4. Measurable disease with at least one lesion that can be accurately measured in at least one dimension (longest dimension recorded). Each lesion must be > 20 mm when measured by conventional techniques, including palpation, plain x-ray, CT and MRI, or > 10 mm when measured by spiral CT. OR Clinically or radiologically detectable disease (ascites, peritoneal deposits, mesenteric thickening or lesions that do not fulfill RECIST for measurable disease). In addition, the subject must have two consecutive rising pretreatment CA-125 levels that are both > 2x the institutional upper limit of normal (ULN) and 40.0 IU/ml taken at least 1 week and nor more than 3 months apart.
5. Platinum-resistant or refractory cancer; subjects must not have had a biologic or chemotherapeutic regimen for treatment of platinum-resistant disease prior to study entry. Subjects with primary platinum-resistant cancer must have had a tumor recurrence within 6 months after completing or while receiving a platinum-containing regimen. These subjects must not have had any other non-platinum-containing regimen. OR Subjects with secondary platinum-resistant cancer may have had any regimen with any response and then have had tumor recurrence within 6 months after completing or while receiving retreatment with a platinum-containing regimen. These subjects must have received only two prior chemotherapeutic regimens. OR Subjects who receive a chemotherapeutic regimen as consolidation after a response to a platinum-containing regimen must have had tumor recurrence within 6 months after completing or while receiving the consolidation regimen.
6. Life expectancy > 12 weeks
7. ECOG performance status 0 or 1
8. Use of an effective means of contraception (for women of childbearing potential)
9. Clinical laboratory test results: Granulocyte count > 1500/µL; Platelet count > 75000/µL; Hemoglobin > 9g/dL (hemoglobin may be supported by transfusion or erythropoietin or other approved hematopoietic growth factors; darbepoetin is permitted); Serum bilirubin < 1.5 the ULN; alkaline phosphatase, AST, and ALT < 2.5 ULN ( AST, ALT < 5.0 ULN for subjects with liver metastasis); Serum creatinine < 1.5 ULN; International normalized ratio (INR) < 1.5 and activated partial thromboplastin time (aPTT) < 1.5 ULN (except for subjects receiving anti-coagulation therapy)

Exclusion Criteria:

1. Prior treatment with gemcitabine
2. Three or more prior chemotherapeutic regimens for the management of primary disease
3. Prior treatment with experimental anti-cancer agents within 4 weeks prior to Day 1 (the day the first study treatment infusions are administered)
4. History or clinical evidence of central nervous system or brain metastases
5. Prior treatment with Avastin or other anti-angiogenic agent
6. Uncontrolled hypercalcemia ( >11.5 mg/dL)
7. History of other malignancies within 5 years of Day 1, except for adequately treated carcinoma in situ of the cervix, ductal carcinoma in situ (DCIS) of breast, basal or squamous cell skin cancer
8. History of serious systemic disease, unstable angina, myocardial infarction, stroke, transient ischemic attack,, symptoms of CHF, or unstable symptomatic arrhythmia requiring medication (subjects with chronic atrial arrhythmia, i.e., atrial fibrillation, paroxysmal supraventricular tachycardia, are eligible) within 6 months prior to Day 1 of treatment
9. Known HIV infection
10. Pregnancy or lactation
11. Major surgery, open biopsy, or significant traumatic injury within 4 weeks prior to Day 1 of treatment, or anticipation of need for major surgical procedure during the course of the study
12. Inability to comply with study and follow-up procedures
13. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the subject at high risk from treatment complications
14. Life expectancy of less than 12 weeks
15. Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study
16. Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
17. Any prior history of hypertensive crisis or hypertensive encephalopathy
18. New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix E)
19. Known CNS disease
20. Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
21. Symptomatic peripheral vascular disease
22. Evidence of bleeding diathesis or coagulopathy
23. Any patient that the clinician considers at risk for possible GI perforation. This includes patients with clinical symptoms or signs of GI obstruction or who require parenteral nutrition, parenteral hydration, or tube feeding, and patients with evidence of free air not explained by paracentesis or recent surgical procedure.
24. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
25. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
26. Serious, non-healing wound, ulcer, or bone fracture
27. Proteinuria at screening as demonstrated by either Urine protein:creatinine (UPC) ratio ≥ 1.0 at screening OR Urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
28. Known hypersensitivity to any component of bevacizumab
29. Pregnant (positive pregnancy test) or lactating. Use of effective means of contraception (men and women) in subjects of child-bearing potential

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  The primary outcome measure is progression-free survival. Disease status and response rates will be determined by investigator assessment using RECIST or CA-125 changes (subjects with nonmeasurable disease only)

SECONDARY OUTCOMES:
Safety and tolerability of bevacizumab in combination with gemcitabine will be assessed. | 2 years
  The safety and tolerability of bevacizumab in combination with gemcitabine will be assessed using the following measures:
  - Incidence, nature, severity, and relatedness of adverse events graded according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE, Version 3.0)

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila Makhija, MD, Principal Investigator — Emory University